CLINICAL TRIAL: NCT05530980
Title: Developing a Lifestyle Intervention to Reduce Body Weight for Obese African American Men Living in the Rural South
Brief Title: "GameDay Ready": Evaluating a Behavioral Weight Management Program for Black Men Living in the Rural South
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Demetrius Abshire, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00116611; K23MD013899 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Physical Inactivity; Diet, Healthy
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GameDay Ready Program (Experimental): The GameDay Ready Program is a 12-week, football-themed, behavioral weight management intervention that promotes gradual increases in physical activity, reductions in sedentary time, and improvements in dietary habits through education, self-monitoring of physical activity and diet, personalized goal setting, group-based competition, social support, identifying and overcoming barriers, and including physical activity as a substantial component of meeting sessions. The program is sensitive to unique cultural influences surrounding gender, race, and rurality; and issues related to motivation are threaded throughout the program.
  Interventions: Behavioral: GameDay Ready Program

INTERVENTIONS:
Behavioral: GameDay Ready Program — GameDay Ready is a 12-week, group-based behavioral weight management program in which participants will meet in-person once per week at a publicly accessible walking track. Each weekly session will be led by a trained facilitator and will include a brief educational component, participant updates on progress, group discussions about overcoming barriers, supervised competitive physical activities, and goal setting for the upcoming week. Educational content will be reinforced and social support will be provided during warmup and cool down walks. Participants will be asked to set behavioral goals toward increasing physical activity and improving dietary habits and will be provided resources to self-monitor their activity, dietary intake, and weight.

SUMMARY:
The primary objective of this study is to test the feasibility and acceptability of a 12-week behavioral weight management intervention adapted for Black men living in the rural South. The intervention is guided by Self-Determination Theory of Motivation, Social Cognitive Theory, and Ecological Systems Theory. Key aspects of the intervention include a football-themed curriculum, facilitator and peer concordance to the extent possible (ie., similarly aged Black men), an emphasis on male-specific health concerns, group-based competition at multiple levels of the intervention (e.g., during in-person physical activity sessions and for achieving behavioral goals), a limited educational component, and physical activity being a substantial component of meeting sessions.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American or Black American male
* BMI 27kg/m^2 to 50kg/m^2 (healthcare provider approval required for those with a BMI >45)
* Able to speak and understand English

Exclusion Criteria:

* Positive response to any question on the Physical Activity Readiness Questionnaire (PAR-Q) (Participant may be included if approval is provided and documented by a healthcare provider)
* Currently participating in another weight loss trial or program or have participated in a trial or program within 6 months prior to starting the intervention
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm hg), diabetes, or asthma (Participant may be included if approval is provided and documented by a healthcare provider)
* Pulmonary disease requiring supplemental oxygen or daily use of short-acting bronchodilators
* Any musculoskeletal condition that would preclude meeting recommended levels of moderate-to-vigorous physical activity
* Within 30 days prior to participating in the intervention, have taken prescription or nonprescription medications, herbals, or supplements for weight loss
* On special diet for a serious health condition (does not include general dietary advice from a healthcare provider for common risk factors such as hypertension, diabetes, or hyperlipidemia)
* Major surgery in the past 6 months
* Have undergone weight loss surgery or considering surgery
* Have been treated for cancer in the past 12 months (other than non-melanoma skin cancer)
* Weight loss ≥5% during the past 6 months
* Any other perceived physical or mental health-related condition that would preclude participating in a behavioral program designed to promote weight loss
* Intending to move within 6 months

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demetrius A Abshire, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon reasonable request.

RESULTS

PARTICIPANT FLOW:
Groups:
- GameDay Ready Intervention: The GameDay Ready Program is a 12-week, football-themed, behavioral weight management intervention that promotes gradual increases in physical activity, reductions in sedentary time, and improvements in dietary habits through education, self-monitoring of physical activity and diet, personalized goal setting, group-based competition, social support, identifying and overcoming barriers, and including physical activity as a substantial component of meeting sessions. The program is sensitive to unique cultural influences surrounding gender, race, and rurality; and issues related to motivation are threaded throughout the program.
Period: Overall Study
Arm/Group | GameDay Ready Intervention
Started | 7
Completed | 4
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | GameDay Ready Intervention
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Study Interest
Description: Number of people expressing interest in the study
Time Frame: Up to week 1
Population: Overall number of participants analyzed represents number of participants screened for study interest prior to enrollment.
Measure: Number; unit: Number of people
Arm/Group | GameDay Ready Program
Number analyzed (Participants) | 91
Number of people | 91

2. Primary Outcome: Eligibility
Description: Number of men who express interest in the study and are eligible.
Time Frame: Up to week 1
Measure: Number; unit: number of people
Arm/Group | GameDay Ready Program
Number analyzed (Participants) | 91
number of people | 14

3. Primary Outcome: Time to Enroll
Description: Length of time needed to enroll the desired sample size (length of time reflects when recruitment was initiated until study launch)
Time Frame: Up to week 1
Population: Overall number of participants analyzed reflects the number of participants who enrolled in the study.
Measure: Number; unit: months
Arm/Group | GameDay Ready Program
Number analyzed (Participants) | 7
months | 5

4. Primary Outcome: Attendance
Description: Number and proportion of enrolled men who attend each intervention session and total number of sessions. Percentage of sessions attended calculated as the total number of sessions attended divided by total number of sessions offered.
Time Frame: Baseline to 3 months
Population: Of the 7 participants who were enrolled in the study, one did not attend any session. One enrolled participant only attended the first session.
Measure: Number; unit: percentage of sessions attended
Units Other Than Participants: Sessions
Arm/Group | GameDay Ready Intervention
Number analyzed (Participants) | 7
Number analyzed (Sessions) | 12
percentage of sessions attended
  Percentage of sessions attended based on 7 enrolled participants. | 49
  Percentage of sessions attended excluding one participant who attended 0 sessions.: number analyzed (Participants) | 6
  Percentage of sessions attended excluding one participant who attended 0 sessions. | 57
  Percentage of sessions attended excluding participants who attended 0 or just 1 session.: number analyzed (Participants) | 5
  Percentage of sessions attended excluding participants who attended 0 or just 1 session. | 67

5. Primary Outcome: Attrition
Description: Number and percentage of enrolled men who withdraw from the study
Time Frame: Baseline to 3 and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GameDay Ready Intervention
Number analyzed (Participants) | 7
Participants
  Number of enrolled participants remaining in study at 3 months. | 5
  Number of enrolled participants remaining in study at 6 months. | 4

6. Secondary Outcome: Change in Weight
Description: Participant body weight measured using a portable, professional-grade scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Body Mass Index
Description: Weight in kilograms divided by height in meters squared
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in Waist Circumference
Description: Measured using an anthropometric measuring tape
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Blood Pressure
Description: Systolic and diastolic blood pressure measured using an a portable automatic monitor
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in Moderate-to-vigorous Physical Activity
Description: Average minutes of moderate-to-vigorous physical activity measured over 7 consecutive days using an accelerometer
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Dietary Intake
Description: Caloric intake, saturated fat intake, fruit and vegetable intake measured using 3-day 24 hour dietary recalls
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

12. Secondary Outcome: Social Support for Diet and Physical Activity
Description: Measured using validated scales developed by Sallis et al.
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

13. Secondary Outcome: Environmental Support for Physical Activity
Description: Measured using the 33-item Rural Active Living Perceived Environmental Support Scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

14. Secondary Outcome: Motivation for Weight Loss
Description: Measured using an 8-item Weight Control Motivation Scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

15. Secondary Outcome: Motivation for Healthy Eating
Description: Measured using a 15-item scale of the Treatment Self-Regulation Questionnaire
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

16. Secondary Outcome: Motivation for Physical Activity
Description: Measured using the 24-item Motivation for Exercise Scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

17. Secondary Outcome: Self-efficacy for Exercise
Description: Measured using a 16-item Self-Efficacy for Exercise Scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

18. Secondary Outcome: Neighborhood Surroundings
Description: Measured using the neighborhood surroundings subscale of the Neighborhood Environment Walkability Scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

19. Secondary Outcome: Neighborhood Safety
Description: Measured using the neighborhood safety subscale of the Neighborhood Environment Walkability Scale
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

20. Secondary Outcome: Relatedness to Others in Physical Activity
Description: Measured using a 6-item scale developed by Wilson & Bengoechea
Time Frame: Change from baseline to 3 and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | GameDay Ready Intervention
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT05530980/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT05530980/SAP_001.pdf